CLINICAL TRIAL: NCT03482284
Title: Exploratory Study on the Modulation of Endotoxemia and Metabolic Parameters: Role of Macronutrients
Brief Title: Effect of Monosaccharides on Intestinal Barrier Function
Acronym: ENDO-META
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Ina Bergheim (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Ina Bergheim, Prof. Dr., University of Vienna
Organization: University of Vienna (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UVienna18
Record Dates: First submitted 2018-03-20; First posted 2018-03-29 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Dietary Habits; Endotoxemia
MeSH Terms: conditions — Feeding Behavior; Endotoxemia | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: All participants receive all interventional diets.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monosaccharide 1 (Experimental): Participants receive standardized meals with a defined amount of monosaccharide 1.
  Interventions: Other: Dietary Intervention
- Monosaccharide 2 (Experimental): Participants receive standardized meals with a defined amount of monosaccharide 2.
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — Participants receive different monosaccharides for a defined number of days.

SUMMARY:
The aim of the present study is to determine the effect of monosaccharides on intestinal barrier function in healthy subjects.

DETAILED DESCRIPTION:
In the intervention study normal weight participants will receive defined amounts of monosaccharides for several days. Before and after intervention parameters of intestinal barrier function will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* BMI <25 kg/m2
* no kown history of metabolic disorders or fatty liver

Exclusion Criteria:

* food allergies or intolerances (esp. fructose intolerance and malabsorption)
* renal insufficiency
* chronic disease of the gastrointestinal tract
* taking drugs affecting lipid or glucose metabolism

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2017-09-09 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Changes in parameters of intestinal barrier function | 1 week
  Changes in endotoxin plasma levels

SECONDARY OUTCOMES:
Changes in blood pressure | 1 week
  Changes in systolic and diastolic blood pressure
Changes in markers for glucose metabolism | 1 week
  Changes in fasting glucose and fasting insulin levels
Changes in blood lipid levels | 1 week
  Changes in triglyceride levels
Changes in Uric Acid levels | 1 week
  Changes in Uric Acid blood levels

IPD SHARING:
Plan to Share IPD: No